CLINICAL TRIAL: NCT06929845
Title: Organoid Models of Hepatocellular Carcinoma to Test Treatment Efficacy, Exploring Correlations With Tumor Microenvironment and Gut-liver-tumor Axis.
Brief Title: Organoid Models of Hepatocellular Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6845
Record Dates: First submitted 2024-07-16; First posted 2025-04-16 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-03

CONDITIONS: Hepatocellular Carcinoma; Organoids; Gut Microbiota; Tumor Microenvironment; System Disorders, Digestive; Surgery
MeSH Terms: conditions — Carcinoma, Hepatocellular; Digestive System Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HCC organoid models development (Experimental): The aim of the present project is to develop a HCC organoid model that closely resembles the in vivo immunological microenvironment, including the contribution of the gut-liver axis. These reconstituted HCC models will then allow us to test tumor sensitiv
  Interventions: Procedure: organoids models

INTERVENTIONS:
Procedure: organoids models — Enrolled patients will undergo liver biopsy with sampling of tumor tissue and adjacent nontumor liver parenchyma. Alternatively, patients who are candidates for surgical resection of HCC will be enrolled. The tumor tissue obtained will be used partly for histological confirmation of HCC and then included in kerosene, partly used for organoid construction, and the nontumor tissue will be used solely for organoids. Genomic and transcriptomic changes resulting from the integration of PDO of HCC with the gut microbiota and host immune cells derived from the patient will be evaluated. In addition, PDOs from HCC will be tested for the efficacy of systemic therapies (ICI and TKI) and understand possible modifying co-factors.

SUMMARY:
A promising tool to elucidate the molecular characteristics of HCC are patient-derived organoids (PDOs), three-dimensional cultures of cells that self-organise according to tissue-specific patterns and can be used to test the susceptibility of a specific tumour to anticancer agents. In this study, PDOs for HCC will be developed that closely resemble the tumour microenvironment in vivo and mimic the crosstalk of the gut-liver axis to establish a correlation with patient prognosis and test the efficacy of available systemic therapies.

DETAILED DESCRIPTION:
The objectives of the project will be 1) to develop HCC PDOs from tumour and non-tumour patient liver tissue obtained from surgical specimens or liver biopsies; 2) to evaluate genomic and transcriptomic changes resulting from the integration of HCC PDOs with patient-derived gut microbiota and host immune cells, and to assess the correlation with patient prognosis; 3) to exploit HCC PDOs to test the efficacy of systemic therapies (ICI and TKIs) and to understand possible modifying cofactors.

Researchers with laboratory experience have been recruited who will focus on the construction of PDOs and the analysis of immune-inflammatory pathways. State-of-the-art technologies will be used, in particular next-generation sequencing, flow cytometry, high-throughput genomic and transcriptomic analysis, ultrafiltration, drug screening, multiplex immunoassays and enzyme immunoassays. The project aims to study the mechanisms involved in the modulation of therapeutic efficacy in patients with HCC. Therefore, the experimental model could be a valuable support to be integrated into real clinical practice to maximise therapeutic efficacy through a fully customised strategy.

ELIGIBILITY:
Inclusion Criteria:

* Capacity to express informed consent;
* Age ≥18 years;
* Suspected radiological diagnosis of HCC or diagnosis of HCC with indications for surgical resection.

Exclusion Criteria:

* Age < 18 years;
* Contraindications to liver biopsy (ascites, platelets<50,000, INR>1.7);
* Contraindications to HCC resection surgery;
* Active viral infection;
* Refusal to sign informed consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Organoid model development | 2-18 months
  The primary endpoint of this study is to assess the correlation between the genomic and histological characteristics of patient-derived organoids (PDOs) from hepatocellular carcinoma (HCC) surgical biopsies and clinical outcomes, specifically disease-free survival (DFS) and overall survival (OS).

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Romana Ponziani, PI, Principal Investigator — Fondazione Policlinico A. Gemelli IRCCS, Rome, Largo A. Gemelli, 8
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, UOC CEMAD, Largo A. Gemelli, 8, Roma, Italy